CLINICAL TRIAL: NCT00248573
Title: Mechanisms of Adaptation in Human Short Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas R. Ziegler, MD, Professor of Medicine, Emory University
Other Study IDs: 0299-2004; R03DK067123 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Intestinal biopsy samples

SUMMARY:
This is an observational, natural history trial of mechanisms of gut adaptation in adult short bowel syndrome (SBS). Patients with SBS (< 200 cm small bowel ± colon) will be studied initially 2-9 months after the last small bowel resection and again exactly 6 months after the initial study. GCRC-studies will examine intestinal nutrient absorption, gut barrier functions and gut mucosal biopsy specimens for markers of nutrient transport and cell proliferation and apoptosis.

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is a condition that occurs after massive surgical removal of sections of the small bowel required to treat conditions such as Crohn's disease, lack of adequate blood flow to the intestine, trauma, twisting of the bowel and other disorders. Patients with SBS develop severe diarrhea, weight loss, loss of nutrients in the stool, malnutrition, dehydration and deficiency of specific nutrients. SBS is thus a major cause of intestinal failure in adults and children. SBS has a high rate of death and medical complications and patients experience enormous health care-related costs and decreased quality of life. Patients with SBS often require intravenous feeding [known as parenteral nutrition (PN)] due to chronic malabsorption and malnutrition and also commonly develop infections from intestinal bacteria, suggesting abnormalities in the intestinal "barrier" to bacteria present in the intestine. In animal models of SBS, increased growth of the intestinal lining (mucosa) and improved nutrient absorption occur over time (intestinal adaptation). Although SBS patients commonly exhibit decreased diet-induced diarrhea within the first 2 years after intestinal surgery, very little is known about how the intestinal mucosa adapts in patients with SBS. The proposed pilot study will be the first comprehensive study of serial changes in gut mucosal structure and function in the early period (2-30 months) of SBS in humans. Our Specific Aims are designed to determine: 1) whether the residual small bowel and colonic mucosa in SBS patients exhibits adaptive growth, with concomitantly improved nutrient absorption and gut barrier function; 2) The underlying mechanisms of early gut adaptation in human SBS, by evaluating changes in mucosal cell growth and production of key molecules that are responsible for nutrient transport/absorption and gut barrier function; and 3) The utility of plasma citrulline concentrations and serum flagellin antibody titers as markers for human intestinal absorptive capacity and gut barrier function, respectively. Our research will provide important and new information on the natural history and underlying causes of early intestinal adaptation in man. This information will be valuable in the design of future therapeutic studies in patients with SBS that hold promise for improving the rehabilitation of these individuals.

ELIGIBILITY:
Inclusion Criteria: 1) Adult male or female with less than 200 small bowel remaining after latest small bowel resection (SBR); 2) Subject able to enter the study within 2-24 months of latest SBR; 3) Age 18-75 years; 4) Body mass index (BMI) ≥ 17 kg/m2; 5) Subject is living at home, clinically stable and expected to survive at least one year; 6) Subject able to take some oral solid diet and oral medications; 7) Intact stomach and duodenum and at least 30 cm of in-continuity jejunum and/or ileum (presence of residual colon is not a specific eligibility criterion); 8) Accurate records available on residual small bowel/colonic length (accurate tape measurement in operation room or small bowel follow-through performed within 3 months of entry); 9) Subject has the ability to understand the requirements of the study, provide written informed consent and agrees to participate in all GCRC assessments.

-

Exclusion Criteria: 1) Evidence of active malignancy during the past 5 years (with the exception of non-metastatic skin cancer; 2) Evidence of uncontrolled hypertension, congestive heart failure, myocardial infarction or angina; 3) History or evidence of stroke or clinically serious neurologic dysfunction since last SBR; 4) Evidence of acute infectious illness requiring hospitalization within the previous 4 weeks; 5) History of steroid-or oxygen-dependent lung disease; 6) History of mental deficiency, alcoholism, or other substance abuse problems; 7) Pregnancy or lactation ; 8) Evidence of worsening of Crohn's disease within 2 months prior to study (i.e. worsening diarrhea, new abdominal pain, rectal bleeding, and, when clinically applicable, abnormal radiographic and/or endoscopic findings); 9) Condition requiring daily systemic corticosteroids exceeding a dose equivalent to 10 mg/d of prednisone or significant immunosuppressant therapy (with the exception of Crohn´s disease); 11) Subject has received glutamine or growth hormone within 2 months prior to study.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1) Adults aged 18-75 with less than 200cm small bowel remaining after latest(SBR); 2) Subject able to enter the study within 2-24 months of latest SBR; 3)(BMI) ≥ 17 kg/m2; 4) Subject is living at home, clinically stable and expected to survive at least one year; 5) Subject able to take some oral solid diet and oral medications; 6) Intact stomach and duodenum and at least 30 cm of in-continuity jejunum and/or ileum (presence of residual colon is not a specific eligibility criterion); 7) Accurate records available on residual small bowel/colonic length (accurate tape measurement in operation room or small bowel follow-through performed within 3 months of entry); 8) Subject has the ability to understand the requirements of the study, provide written informed consent and agrees to participate in all assessments.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2004-10; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
intestinal gene expression | 2011-2012

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania